CLINICAL TRIAL: NCT00325091
Title: Long-Term Motor Learning in Focal Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060161; 06-N-0161
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-01-06

CONDITIONS: Focal Hand Dystonia
Keywords: Writer's Cramp; Electroencephalogram (EEG); Transcranial Magnetic Stimulation (TMS); Fine Motor Skills; Focal Hand Dystonia; Writer Cramp; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia, Focal, Task-Specific; Dystonic Disorders

SUMMARY:
This study will examine the effects of long-term practice of repeated finger movements in people with focal hand dystonia, as compared with healthy volunteers. Patients with dystonia have muscle spasms that cause abnormal postures while trying to perform a movement. In focal dystonia, just one part of the body, such as the hand, neck or face, is involved.

Right-handed healthy volunteers and patients with focal hand dystonia of the right hand 18 years of age and older may be eligible for this study. Candidates are screened with a medical history and neurological and physical examination.

Participants are trained daily for 11 days (excluding weekends) at the NIH and are asked to continue with daily 15 minutes of practice over a 12-week period to perform sequential finger movement task (key presses) with their left hand. They practice initially at NIH and then at home. At each clinic visit, their learning of the motor skill is assessed by recording their performance of 20 consecutive trials of the eight sequences (a total of 160 key presses) in the task.

To evaluate long-term motor learning of the sequential movements, participants are asked to do different task tests at Day 2, Week 4 and Week 12. Brain wave activity, and brain excitability are also measured during these days. In one task, they see a random series of letters on a screen during the sequential finger movements and are asked to say the number of times they see a specific letter. In another task, they are asked to focus on each specific movement while performing the sequential finger movements. During each visit, they are questioned and evaluated for the development of any abnormal movements that may be suggestive of early dystonia.

All participants have an electroencephalogram (EEG) and transcranial magnetic stimulation (TMS) at Day 1, and Day 2 and at Week 4 and Week 12 to evaluate brain activity. For the EEG, electrodes are placed on the subject's scalp and the electrical activity of the brain is recorded while the subject performs the sequence of finger movements. For TMS, a wire coil is held on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The effect of TMS on the muscles is detected with small electrodes taped to the skin of the subject's arms or legs.

...

DETAILED DESCRIPTION:
OBJECTIVE:

The overall goal of this proposal is to provide new insights into long-term motor learning by studying patients with focal hand dystonia (FHD) and healthy controls. Long-term motor learning has never been studied in FHD patients. Our central hypothesis is that dystonia is caused by abnormal long-term motor learning. Specifically, the aims of this study are:

1. To show that FHD patients have abnormal motor learning, and in particular, have slower motor skill acquisition compared to healthy controls.
2. To show that FHD patients have difficulty in performing newly acquired motor skills automatically.
3. To study brain dynamics (i.e. cortico-cortical connectivity and motor cortex excitability) in FHD patients and healthy controls while learning a sequence of finger movements over a 3-month period of time.

STUDY POPULATION:

We will follow 10 patients with FHD affecting their dominant hand and 10 healthy volunteers.

DESIGN:

We have devised this case-control experimental study to evaluate the long-term learning of sequential finger movements in FHD patients and healthy controls. We will study FHD patients and healthy volunteers for 12 weeks as they learn a 4 finger sequence of eight key presses with their left hand using a metronome to mark the rhythm. All subjects will be right-handed and age-matched. They will be asked to practice this sequence of 8 key presses daily for 30 minutes for the first week and then for 15 minutes for the remainder of the study. For the first 3 weeks of the study, subjects will come to the Clinical Center (CC) 10 times at regular intervals based on their availability. They will practice daily at the CC or at home during this period. They will then come to the CC every 2 weeks (plus or minus 3 days) for the remainder of the study while practicing daily for 15 minutes. At each visit, learning will be assessed by measuring the sequence error rates (SER) and variability in the interval between key presses. All subjects will be asked to keep a log of daily practice during the 12 weeks. At each visit patients will be carefully questioned and evaluated for the development of abnormal movement patterns suggestive of early dystonia.

OUTCOME MEASURES:

The primary outcome of this study will be to measure the SER at baseline, week 4 and week 12 using 20 consecutive trials of the 8 sequences. We will measure multiple secondary outcomes: (a) variability in the interval between key presses; (b) automaticity of the movement evaluated by a dual task; (c) constrained action evaluated by a thinking task; (d) transcranial magnetic stimulation (TMS) and electroencephalography (EEG) studies to explore changes in brain physiology.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers:

* Age 18 years and older
* Right-hand dominant (Edinburgh Handedness Quotient greater than 60)
* Able to provide consent for the protocol

Patients:

* Age 18 years and older
* Right hand dominant (Edinburgh Handedness Quotient greater than 60)
* Idiopathic focal hand dystonia in right hand
* Able to provide consent for the protocol

EXCLUSION CRITERIA:

* Subjects with other medical, surgical, neurologic or psychiatric conditions
* If participants are taking certain centrally acting medications (like antidepressants, anxiolytics/neuroleptics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines) may not be eligible to participate in this study.
* The presence of a cardiac pacemaker, an implanted medical pump, a metal plate or metal object in skull or eye is contraindications for TMS application.
* Patients with seizure disorder or epilepsy
* Subjects without the capacity to give informed consent
* If participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as excessive fatigue, general frailty, or excessive apprehension

Patients:

* Subjects with any abnormal findings on neurological examination (except right hand), and general physical examination
* Secondary hand dystonia

Healthy volunteers:

* Subjects with any abnormal findings on neurological examination and general physical examination
* Subjects who have learned to play the piano or any other keyboard instrument in the past.
* Subjects who have jobs or are involved in daily activities that demand skilled, fine-finger movements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-05-09; Study Completion 2014-01-06

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agostino R, Berardelli A, Formica A, Accornero N, Manfredi M. Sequential arm movements in patients with Parkinson's disease, Huntington's disease and dystonia. Brain. 1992 Oct;115 ( Pt 5):1481-95. doi: 10.1093/brain/115.5.1481. PMID 1422799
- [Background] Andres FG, Mima T, Schulman AE, Dichgans J, Hallett M, Gerloff C. Functional coupling of human cortical sensorimotor areas during bimanual skill acquisition. Brain. 1999 May;122 ( Pt 5):855-70. doi: 10.1093/brain/122.5.855. PMID 10355671
- [Background] Byl NN, Merzenich MM, Jenkins WM. A primate genesis model of focal dystonia and repetitive strain injury: I. Learning-induced dedifferentiation of the representation of the hand in the primary somatosensory cortex in adult monkeys. Neurology. 1996 Aug;47(2):508-20. doi: 10.1212/wnl.47.2.508. PMID 8757029